CLINICAL TRIAL: NCT01502735
Title: A Phase 1 Trial of the Walter Reed Army Institute of Research (WRAIR) Dengue Virus Serotype-1 Purified Inactivated Vaccine (DENV-1 PIV) in Flavivirus Antibody Naïve Adults
Brief Title: Safety Study of a Vaccine (DENV-1 PIV) to Prevent Dengue Disease
Acronym: DENV-1 PIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-10-0003; WRAIR IRB Protocol # 1856 (Other: WRAIR); HSRRB Protocol #: A-17104 (Other: HSRRB); IND 14338 (Other: FDA)
Record Dates: First submitted 2011-12-16; First posted 2012-01-02 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Dengue Fever
Keywords: dengue; dengue fever; monovalent dengue vaccine
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DENV-1 PIV (high dose) (Experimental)
  Interventions: Biological: DENV-1 PIV, 5 µg
- DENV-1 PIV (low dose) (Experimental)
  Interventions: Biological: DENV-1 PIV, 2.5 µg

INTERVENTIONS:
Biological: DENV-1 PIV, 2.5 µg — 2.5 µg Purified Inactivated Virus (PIV) in a volume of 0.5 mL administered via intramuscular injection on Study Days 0, and 28 (±4 days)
  Arms: DENV-1 PIV (low dose)
Biological: DENV-1 PIV, 5 µg — 5 µg Purified Inactivated Virus (PIV) in a volume of 0.5 mL administered via intramuscular injection on Study Days 0, and 28 (±4 days)
  Arms: DENV-1 PIV (high dose)

SUMMARY:
This is a phase 1 study to evaluate the safety of a vaccine (DENV-1 PIV) for the prevention of dengue fever.

DETAILED DESCRIPTION:
DENV infections can cause self-limited but incapacitating acute illness lasting four to seven days. The illness is characterized by fever, headache, severe pain in muscles, joints, pain behind the eyes, and a rash. DENV infection can be complicated by the development of hemorrhagic fever (DHF) or shock syndrome (DSS), which is manifested by plasma leakage and a bleeding diathesis or frank hemorrhage. DHF is fatal in at least 0.5% of pediatric cases but rarely in adults. People, particularly children, living in hyper-endemic areas who have antibodies from an earlier dengue infection with one serotype are at increased risk for DHF if subsequently infected by another dengue virus serotype.

Currently, no specific anti-viral therapy exists. Therapy is largely supportive. Mosquito control has failed to prevent dengue transmission; therefore, prevention of dengue through vaccination is an important objective of the World Health Organization (WHO) and many national governments, including the United States.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years of age or the legal age of consent (whichever is greater) to 50 (inclusive) years of age
* Negative screening laboratory test against dengue, Japanese Encephalitis, West Nile, and Yellow Fever viruses
* Healthy
* All subjects must agree to use contraception or to abstain from sex from enrollment through trial completion
* Able to provide informed consent and able to be followed throughout the trial period

Exclusion Criteria:

* History of Flavivirus infection or history of Flavivirus vaccine (experimental or licensed product) including Japanese encephalitis, West Nile virus, Yellow fever, and dengue
* Have a known or suspected hypersensitivity or adverse reaction to vaccines
* Have received a live-attenuated vaccine within 42 days prior to the initial injection on Day 0 or a subunit or killed vaccine within 30 days of the initial injection on Day 0
* Are pregnant or breastfeeding
* Known HIV, Hepatitis B and/or Hepatitis C infection
* Have any acute illness, including an oral body temperature greater than 100.4°F at the day of vaccination
* Have any occupational, social, or medical concerns that would impact subject safety, interfere with protocol adherence, or affect a subject's ability to give informed consent
* Have been using immunomodulatory therapy (use of systemic corticosteroids or chemotherapeutics that may influence antibody development) within the past 6 months; medications or nutritional supplements known to or which potentially could affect organ function within 30 days prior to the initial injection
* Have received an investigational drug or vaccine or participated in a drug product or vaccine study within a period of 30 days prior to Day 0
* Have received or donated blood or plasma within 90 days of Day 0 (or plan on receiving or donating blood or plasma during the study)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects with solicited adverse events (AEs) from study day 0 to 90 | Up to 90 days
Number of subjects with unsolicited AEs from study day 0 to 90 | Up to 90 days
Number of subjects who experience serious adverse events (SAEs) during the study period | Up to 360 Days

SECONDARY OUTCOMES:
Number of subjects with a change in geometric mean titer of neutralizing antibody to DENV types 1,2,3, and 4 | Up to Day 28
Number of subjects with a change in geometric mean titer of neutralizing antibody to DENV types 1,2,3, and 4 | Up to Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Thomas, MD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- WRAIR, Clinical Trials Center (CTC), Silver Spring, Maryland, United States